CLINICAL TRIAL: NCT06925880
Title: Efficacy of Supplementation With Micronized Creatine Monohydrate in the Recovery of Muscle Mass, Muscle Strength and Functional Capacity in Older Adults Operated on for Total Knee Arthroplasty: Randomized Clinical Trial
Brief Title: Effect of Micronized Creatine Monohydrate on Muscle Mass, Strength and Performance in Older Adults Submitted to Total Knee Arthroplasty
Acronym: CREAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Maresme (Other)
Collaborators: Fundació Privada Salut del Consorci Sanitari del Maresme (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIm CSdM 24/25
Record Dates: First submitted 2025-03-27; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia in Elderly; Frailty at Older Adults; Functional Capacity; Creatine Supplementation; Arthroplasties, Knee Replacement; Physical Performance
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CREATINE (Experimental): The intervention will consist of daily supplementation with micronized creatine monohydrate for 12 weeks. The intervention will start at the time of hospital discharge with a loading dose of 20g/day for 1 week. Subsequently, a maintenance dose of 5g/day will be continued for 11 weeks.
  Interventions: Dietary Supplement: Creatine Monohydrate
- PLACEBO (Placebo Comparator): The control group will follow the same rehabilitation regimen as the intervention group and will receive a placebo. It will start at the time of hospital discharge with a loading dose of 20g/day for 1 week. Subsequently, a maintenance dose of 5g/day will be continued for 11 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — The intervention will consist of daily supplementation with micronized creatine monohydrate (FullGas Sport Creatine 200 mesh) for 12 weeks. The intervention will start at the time of hospital discharge with a loading dose of 20g/day for 1 week, divided into 4 intakes of 5g to favor digestive tolerance (breakfast, lunch, snack and dinner). Subsequently, a maintenance dose of 5g/day will be continued for 11 weeks (breakfast). Creatine should be consumed with food to improve its absorption.
  Arms: CREATINE
Other: Placebo — The control group will follow the same rehabilitation regimen as the intervention group and will receive a placebo with FullGas Sport microcrystalline cellulose. Its physical and organoleptic characteristics are the same as micronized creatine monohydrate. The dosage will be the same as that indicated for the study intervention: it will start at the time of hospital discharge with a loading dose of 20g/day for 1 week, divided into 4 intakes of 5g to favor digestive tolerance (breakfast, lunch, snack and dinner). Subsequently, a maintenance dose of 5g/day will be continued for 11 weeks (breakfast).
  Arms: PLACEBO

SUMMARY:
Double-blind randomized placebo-controlled clinical trial with two parallel arms. The main objective is to evaluate the efficacy and safety of creatine supplementation in older adults who have been operated on for total knee arthroplasty and undergoing a usual rehabilitation program. The intervention will consist of daily creatine monohydrate supplementation for 12 weeks. The intervention will start after surgery with a loading dose of 20g/day for 1 week and then continue with a maintenance dose of 5g/day for 11 weeks.

Main outcome mesures included muscle mass, muscle strenght, sarcopenia, frailty, functional capacity and physical performance and will be assessed at baseline, 3 and 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Persons 65 years of age or older who have been operated on for the first time for total knee arthroplasty,
* who are undergoing an outpatient rehabilitation program according to standard clinical practice,
* who sign the informed consent form.

Exclusion Criteria:

* Chronic renal disease at stage G3b or higher or glomerular filtration rate <30 ml/min/1.73m2.
* Hepatic insufficiency, cirrhosis.
* Neuromuscular and neurodegenerative diseases (amyotrophic lateral sclerosis, multiple sclerosis, muscular dystrophy, myasthenia gravis, Parkinson's disease, etc.).
* Severe or very severe chronic obstructive pulmonary disease (COPD) (GOLD III-IV).
* Moderate or severe chronic heart failure (NYHA 3-4).
* Central sensitivity syndrome (fibromyalgia and chronic fatigue syndrome).
* Moderate or severe cognitive impairment (GDS≥4).
* Moderate-severe dependence for basic activities of daily living (preintervention Barthel index <60 points).
* Hemiparesis, amputation or malformation of any limb.
* Consumption of creatine monohydrate supplements in the last 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2025-04-22 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in muscle mass | Baseline, 3 and 6 months follow-up
  Mesured by Bioimpedance Analysis
Change in Muscle Strenght | Baseline, 3 and 6 months follow-up
  Handgrip mesured by Jamar Dynamometer
Change in the prevalence of Sarcopenia | Baseline, 3 and 6 months follow-up
  Mesured by EWGSOP2 criteria
Change in Functional Capacity | Baseline, 3 and 6 months follow-up
  Mesured by Barthel score
Changes in Performance | Baseline, 3 and 6 months follow-up
  Mesured by Timed Up and Go Test (seconds)
Changes in Physical Performance | Baseline, 3 and 6 months follow-up
  Mesured by Short Physical Performance Batery (SPPB)
Changes in aerobic capacity | Baseline, 3 and 6 months follow-up
  Mesured by 6 minutes Walking Test (meters)
Changes in Walking Speed | Baseline, 3 and 6 months follow-up
  Mesured by Gaid Speed
Number of Advers Health Events | Baseline, 3 and 6 months follow-up
  Register of advers health events

SECONDARY OUTCOMES:
Change in Frailty status | Baseline, 3 and 6 months follow-up
  Mesured by Linda Fried criteria (0 positive criteria: robust, 1-2: pre-frail positive criteria, 3 or more positive criteria: frail)
Arthroscopy complications | Baseline, 3 and 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jéssica Martínez Rodríguez, Principal Investigator — Consorci Sanitari del Maresme; Mateu Serra-Prat, PhD, Study Director — Consorci Sanitari del Maresme

IPD SHARING:
Plan to Share IPD: No